CLINICAL TRIAL: NCT01070290
Title: A Randomized Phase 2 Study of ARQ 197 Versus Investigator's Choice of Second-Line Chemotherapy in Patients With Locally Advanced or Metastatic Gastric Cancer Who Have Progressive Neoplastic Disease Following Treatment With One Prior Chemotherapy Regimen
Brief Title: A Study of ARQ 197 Versus Investigator's Choice of Second-Line Chemotherapy in Patients With Locally Advanced or Metastatic Gastric Cancer Who Have Progressive Neoplastic Disease Following Treatment With One Prior Chemotherapy Regimen
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-206
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Gastric Cancer
Keywords: gastric carcinoma; Locally Advanced or Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — ARQ 197; Oxaliplatin; Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ARQ 197
  Interventions: Drug: ARQ 197
- 2 (Active Comparator): Investigator's choice of oxaliplatin, capecitabine or irinotecan
  Interventions: Drug: Oxaliplatin, capecitabine or irinotecan

INTERVENTIONS:
Drug: ARQ 197 — 120 mg capsule administered twice daily
  Arms: 1
Drug: Oxaliplatin, capecitabine or irinotecan — Investigator's choice or oxaliplatin, capecitabine or irinotecan
  Arms: 2

SUMMARY:
This will be a multi-center, open-label randomized phase 2 study designed to evaluate the progression free survival (PFS) of patients with advanced gastric cancer following treatment with either ARQ 197 or one of three standard regimens (investigator's choice). Patients with unresectable (locally advanced or metastatic) gastric carcinoma who have progressive neoplastic disease following treatment with a prior regimen consisting of at least two of the drugs 5-FU, cisplatin and docetaxel. The study will also evaluate other efficacy and safety parameters including overall response rate, overall survival and adverse events in the two treatment arms.

DETAILED DESCRIPTION:
This will be a multi-center, open-label randomized phase 2 study designed to evaluate the PFS of ARQ 197 versus investigator's choice of second-line chemotherapy in patients with unresectable (locally advanced or metastatic) gastric carcinoma who have progressive neoplastic disease following treatment with a prior regimen consisting of at least two of the drugs 5-FU, cisplatin and docetaxel. Patients will be randomized to ARQ 197 arm or investigator's choice arm in a 1:1 ratio. The study will also evaluate other efficacy and safety parameters including ORR, OS and adverse events in the two treatment arms.

Patients assigned to the investigator's choice arm may receive any one of the following:

* Oxaliplatin 85 mg/m2 i.v. every two weeks (each cycle = 4 weeks)
* Capecitabine 1250 mg/m2 p.o. twice daily for 14 days followed by 7 days of no therapy every 3 weeks (each cycle = 3 weeks)
* Irinotecan 125 mg/m2 i.v. weekly for 4 weeks followed by 2 weeks of no therapy every 6 weeks (each cycle = 6 weeks) Treatment will continue unless one of the treatment discontinuation criteria is met. Dose reductions should occur based on the current labels for each of the investigator choice agents.

Patients randomly assigned to the ARQ arm will receive 120 mg of ARQ 197 twice daily (240 mg/day) throughout the treatment period. The treatment of ARQ 197 can be continued until unacceptable toxicity, documented progression of disease, or another discontinuation criterion is met. A cycle of ARQ 197 treatment will be defined as 21 days and cycles may be repeated every 3 weeks (21 days) based on toxicity and response.

The assigned treatment should continue until unacceptable toxicity, disease progression (clinical or radiological) or another discontinuation criterion is met.

Tumor evaluations: Tumor evaluations will be performed at 6-week or 8-week intervals. Tumor response will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST).

Progression-free survival: The time of disease progression-free will be calculated from date of randomization until disease progression per RECIST or death due to any cause. Patients who are alive and progression free will be censored at the date of their last tumor evaluation.

Overall response rate: The ORR will be calculated for the intent to treat patient population as the number of patients with a confirmed complete response or partial response divided by the number of randomized patients.

Overall survival: Overall survival time will be calculated from the date of randomization until death due to any cause.

Safety assessments: Data on vital signs, physical examination, adverse events, serum chemistry, hematological laboratory tests, and electrocardiograms will be collected.

Based on the data for irinotecan, it is estimated that the median PFS in the second-line chemotherapy arm will be 4 months. In order to demonstrate an improvement in median PFS to 5.5 months (37.5% improvement, hazard ratio of 0.73) based on a two-sided log rang test, 338 patients (169 per arm) will be required, assuming an 18 month enrollment and a 12 month follow-up, an alpha of 0.05 and 90% power. The sample size assumes a 10% loss to follow-up rate.

A futility analysis will be performed when 33% of the events required for the final analysis have occurred by an Independent Data Monitoring Committee. The futility boundary will be described in the full statistical analysis plan for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent prior to study-specific screening procedures
2. ≥ 18 years old
3. Histologically or cytologically confirmed locally advanced or metastatic unresectable gastric carcinoma
4. Progressive neoplastic disease despite treatment with a regimen consisting of at least two of the following agents given concurrently: 5-FU, cisplatin and docetaxel OR intolerance to such a regimen
5. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
6. Eastern Cooperative Oncology Group performance status 0 to 2
7. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
8. Females of childbearing potential must have a negative serum pregnancy test
9. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN with known metastatic liver disease
10. Total bilirubin ≤ 1.5 × ULN
11. Serum creatinine ≤ 1.5 x ULN
12. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
13. Platelets ≥ 100 x 10^9/L

Exclusion Criteria:

1. Received more than one prior systemic regimen for the treatment of gastric cancer (including chemotherapy, immunotherapy, vaccines, monoclonal antibodies)
2. Known or suspected central nervous system metastases
3. Pregnant or lactating
4. Significant gastrointestinal disorder that, in the opinion of Investigator, could interfere with the absorption of ARQ 197 (e.g. Crohn's disease, ulcerative colitis, extensive gastric resection)
5. Unable or unwilling to swallow ARQ 197 capsules twice daily
6. Any contraindication to treatment with ARQ 197, capecitabine, oxaliplatin or irinotecan
7. Prior treatment with capecitabine, oxaliplatin or irinotecan
8. Any known hypersensitivity to any of the components of ARQ 197, capecitabine, oxaliplatin or irinotecan
9. Treatment with an investigational agent within 30 days of first dose of protocol defined treatments
10. Other malignancies within the last five years, with the exception of adequately treated intraepithelial carcinoma of the cervix uteri, prostate carcinoma with a PSA value < 0.2 ng/ml or basal or squamous cell carcinoma of the skin
11. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation
12. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Compare the progression-free survival (PFS) of ARQ 197 versus investigator's choice of second-line chemotherapy in patients with advanced gastric cancer who have failed first-line treatment.

SECONDARY OUTCOMES:
Compare overall response rate (ORR) of ARQ 197 versus investigator's choice of second-line chemotherapy
Compare 6-month and 1-year overall survival (OS) rates of ARQ 197 versus investigator's choice of second-line chemotherapy
Further characterize the safety profile of ARQ 197